CLINICAL TRIAL: NCT06291350
Title: Characterization of Peroodontal and Intestinal Microbiota in Patients With Gingival Scarring Pemphigoid: a Matched Controlled Study
Brief Title: Peridontal and Intestinal Microbiota in Patients With Gingival Scarring Pemphigoid
Acronym: MICROPC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23-AOI-05
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pemphigoid, Benign Mucous Membrane; Gingivitis Hyperplastic
MeSH Terms: conditions — Pemphigoid, Benign Mucous Membrane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plaque and stool collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MMPg and periodontitis: 15 adult patients with MMPg and periodontitis
  Interventions: Other: Plaque sampling and stool collection; Other: periodontal examination
- no MMPg and periodontitis: 15 adult patients not suffering from MMPg with periodontitis
  Interventions: Other: Plaque sampling and stool collection; Other: periodontal examination
- no MMPg with healthy periodontal conditions: 15 adult patients not suffering from MMPg with healthy periodontal conditions
  Interventions: Other: Plaque sampling and stool collection; Other: periodontal examination

INTERVENTIONS:
Other: Plaque sampling and stool collection — Characterization of the periodontal and digestive microbiota (metagenomic analysis), assessment of clinical attachment loss and alveolysis
Other: periodontal examination — Characterization of the periodontal and digestive microbiota (metagenomic analysis), assessment of clinical attachment loss and alveolysis

SUMMARY:
Patients suffering from Mucous Membrane Pemphigoid with desquamative gingivitis (MMPg) generally present a more degraded periodontal condition compared with controls. Bullous disease could represent a risk factor for plaque-induced periodontal disease, and vice versa.

Indeed, the dysbiotic periodontal microbiota could aggravate the gingival damage specific to MMP, either directly by activating inflammatory pathways, or indirectly by degrading cellular and matrix components. On the other hand, areas of erosive gingiva generated by the autoimmune process could increase the virulent power of periodontal pathobionts, by representing accessible, nutrient-rich connective surfaces. Moreover, in recent years, bacterial studies based on a high-throughput metagenomic approach have suggested the existence of a relationship between the oral and intestinal microbiota in patients with degraded periodontal conditions and suffering from autoimmune inflammatory diseases (inflammatory bowel disease, acute graft-versus-host disease). This relationship can also be envisaged in MMPg patients who meet the conditions that allow this type of pathological process to occur: autoimmune disease; disruption of the gingival epithelial barrier in erosive gingival areas (increasing the risk of antigen exposure); large amounts of thick plaque; degraded periodontal condition with the presence of numerous periodontal pockets from which periodontopathogenic bacteria can translocate intra-tissularly and cause distant adverse consequences.

The main aim of this observational, multicentre, case-control, matched study is to compare the composition of the periodontal microbiota between MMPg patients and control patients (arm 2 and arm 3). The secondary objectives are to compare the composition of periodontal and intestinal microbiota in cases and control patients (arm 2 and arm 3), to compare periodontal microbiota composition in cases and control patients (arm 2) according to periodontitis severity, and to compare gut microbiota composition between cases and control patients (arm 2 and arm3). To date, no such study exists.

ELIGIBILITY:
Inclusion Criteria:

Adults (over 18), non-smokers Arm 1

* MMPg (initial, persistent despite medical treatment, recurrent), periodontitis Arm 2
* non-MMPg, periodontitis, matched to cases on age, gender and severity of periodontitis

Arm 3:

- non-MMPg, healthy periodontal conditions, matched to cases on age and gender

Exclusion Criteria:

* Antibiotic therapy and mechanical periodontal treatment within 3 months prior to study, other chronic general illness of immune or digestive origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: 15 adult patients (over 18 years of age) with CP with erosive gingival expression (CP patients).
  Control group 1: 15 adult patients (over 18 years of age) without CP, matched to cases on age, gender and periodontal conditions.
  Control group 2: 15 adult patients (over 18 years of age) without CP, with healed periodontal conditions, matched to cases on age and gender.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
composition of the periodontal microbiota | at inclusion
  Compare the composition (name and number of bacterial colonies) of the periodontal microbiota between patients with MMPg and periodontitis (cases) and control patients (non-MMPg with case-matched periodontitis or non-MMPg with healthy periodontium)
  Identification and quantification of bacterial populations in the subgingival plaque of cases and controls: global shotgun metagenomic approach, genetic sequencing on a third-generation sequencer

SECONDARY OUTCOMES:
Compare the composition (name and number of bacterial colonies) of periodontal in MMP and control patients (arm 2 and arm 3). | at inclusion
Compare the composition (name and number of bacterial colonies) intestinal microbiota in MMP and control patients (arm 2 and arm 3). | at inclusion
  stool sampling at the patient's home after inclusion
Compare (name and number of bacterial colonies) periodontal microbiota composition in MMP and control patients (arm 2) according to periodontitis severity (non-severe/severe) | at inclusion
Compare (name and number of bacterial colonies) gut microbiota composition between MMP and control patients (arm 2 and arm3) | at inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nice University Hospital, Nice
  - Paris hospital Pitié Salpetrière (APHP), Paris
  - Paris hospital Bretonneau (APHP), Paris

IPD SHARING:
Plan to Share IPD: No